CLINICAL TRIAL: NCT01564680
Title: Intravenous Lornoxicam is More Effective Than Paracetamol as a Supplemental Analgesic After Lower Abdominal Surgery; A Randomized Controlled Trial
Brief Title: Lornoxicam vs. Paracetamol After Lower Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #201021
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Pain
Keywords: Lower abdominal surgery; Paracetamol; Lornoxicam; Morphine
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; lornoxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lornoxicam (Experimental): Lornoxicam 16 mg will be given at skin closure and 8 mg will be given 12 hours postoperatively
  Interventions: Drug: Lornoxicam
- Control (Placebo Comparator): Patients will receive normal saline at skin closure, at 6, 12, 18 hours postoperatively.
  Interventions: Other: placebo
- Paracetamol (Experimental): 1 gm of paracetamol will be given at skin closure, 6, 12, 18 hours postoperatively
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Other: placebo — normal saline
  Other Names: 0.9 N sodium chloride
  Arms: Control
Drug: Paracetamol — IV paracetamol infusion
  Other Names: perfalgan
  Arms: Paracetamol
Drug: Lornoxicam — 16 mg at skin closure and 8 mg 12 hours postoperative
  Other Names: xefo
  Arms: Lornoxicam

SUMMARY:
Background: The aim of this prospective, randomized, double-blind study is to determine the most effective supplemental analgesic, paracetamol or lornoxicam for postoperative pain relief after lower abdominal surgery.

Methods: Sixty patients scheduled for lower abdominal surgery under general anesthesia were randomly allocated to receive either isotonic saline (Control group), intravenous paracetamol 1 g every 6 h (Paracetamol group) or lornoxicam 16 mg then 8 mg after 12 h (Lornoxicam group). Additionally pain was treated postoperatively using morphine patient-controlled analgesia. Postoperative pain scores measured by the verbal pain score (VPS), morphine consumption and the incidence of side effects were measured at 1, 2, 4, 8, 12 and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* lower abdominal surgery

Exclusion Criteria:

* body weight more than 150% of their ideal body weight
* history of significant cardiac, pulmonary, renal, hepatic or hematological disease; chronic drug or alcohol abuse; hypersensitivity to any of the studied drugs; bronchial asthma; gastritis or peptic ulcer; and pregnancy
* patients who received any analgesic drug a day before surgery

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  Postoperative pain scores measured by the verbal pain score (VPS)1, 2, 4, 8, 12 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Morphine consumption | 24 hours
  pain was treated postoperatively using morphine patient-controlled analgesia. Morphine consumption was measured at 1, 2, 4, 8, 12 and 24 hours postoperatively
Incidence of side-effects | 24 hours
  incidence of side effects was measured at 1,2,4,8, 12, 24 hr postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hany A Mowafi, MD, Principal Investigator — UD
Locations (1):
- Dammam University, KFHU, Khobar, EP, Saudi Arabia

REFERENCES:
- [Derived] Mowafi HA, Elmakarim EA, Ismail S, Al-Mahdy M, El-Saflan AE, Elsaid AS. Intravenous lornoxicam is more effective than paracetamol as a supplemental analgesic after lower abdominal surgery: a randomized controlled trial. World J Surg. 2012 Sep;36(9):2039-44. doi: 10.1007/s00268-012-1649-2. PMID 22584689